CLINICAL TRIAL: NCT07007702
Title: Anti-inflammatory Effects and Clinical Efficacy of Topical Thealoz Total Eye Drops in Patients With Chronic Dry Eye Disease and Associated Ocular Surface Inflammation
Brief Title: Anti-inflammatory Effects and Clinical Efficacy of Topical Thealoz Total Eye Drops in Patients With Chronic Dry Eye Disease
Status: Completed | Type: Observational
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Other Study IDs: LT2769-005
Record Dates: First submitted 2025-04-17; First posted 2025-06-06 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Dry Eye Disease (DED)
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Schirmer test strips stored for proteomics and lipidomics analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group receiving T2769
  Interventions: Device: T2769

INTERVENTIONS:
Device: T2769 — Preservative-free combination of trehalose, sodium hyaluronate and N-Acetyl Aspartyl Glutamic Acid

SUMMARY:
The goal of this prospective, open, monocentric study is to evaluate the clinical efficacy of a new preservative-free combination of trehalose, sodium hyaluronate and NAAGA in 30 patients with chronic dry eye disease and associated ocular surface inflammation.

The main question it aims to answer is:

- To assess the improvement of conjunctival hyperemia as well as subjective symptoms in patients with moderate to severe dry eye.

Participants will be asked to use T2769 on a daily basis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Normal ophthalmic findings except dry eye disease
* Chronic dry eye defined as longer than six months since diagnosis
* OSDI ≥ 22
* Conjunctival Hyperemia≥ Grade 3 (Efron Scale)
* Current use of topical lubricants since at least 3 months

Exclusion Criteria:

Ophthalmic exclusion criteria

* Best far corrected visual acuity < 1/10
* Severe Dry Eye associated with:

  * Eyelid malposition
  * Sjogren Syndrome
  * Stevens Johnson Syndrome
  * Corneal dystrophy
  * Ocular neoplasia
  * Filamentous keratitis
  * Corneal neovascularisation
  * Orbital radiotherapy
  * Dry eye related to GVHD
* History of any of the following within last 3 months:
* Systemic treatment of dry eye
* Systemic treatment of MGD
* Isotretinoïde,
* Cyclosporine,
* Tacrolimus, Siromilus, Pimecrolimus
* Punctual plugs
* History of any of the following within previous six months:
* ocular trauma
* ocular infection, Ocular allergy
* History of any of the following within last 12 months:
* inflammatory corneal ulcer
* Herpetic eye infection
* or uveitis
* Ocular surgery

Systemic / non ophthalmic exclusion criteria:

• Known hypersensitivity to any of the components of the medical device under investigation or other study medication

Specific exclusion criteria for women:

* Pregnant or breast-feeding woman.
* Woman of childbearing potential (neither menopausal, nor hysterectomized, nor sterilized) not using effective contraception (i.e. hormonal contraceptives, intra-uterine device, contraceptive implant or condoms)

Exclusion criteria related to general conditions

* Inability of patient to understand the investigation procedures and thus inability to give valid, informed consent.
* Non-compliant patient (e.g. not willing to attend the follow-up visits, way of life interfering with compliance)
* Participation in another clinical study or clinical investigation at the same time as the present investigation
* Participation to the present clinical investigation during the exclusion period of another clinical study
* Patient already included once in this clinical investigation
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 30 patients with moderate to severe dry eye disease and associated inflammation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with Visual Analog Scale (0-10) at week 12 - Descriptive analysis | at week 12
  Scores will be determined using a 100 mm VAS on which 0 means "I do not agree" and 100 means "I totally agree". The following questions will be assessed using VAS:
  "I feel satisfied using this treatment" "With these eye drops, I have a feeling of freshness" "With these eye drops, I have a feeling of relief" "This product contributed to reduce my pain due to eye dryness" "This product is comfortable"
Conjunctival hyperaemia assesment with Efron scale at week 12 | week 12
  Conjunctival hyperemia grading with Photographs (Efron) scale at week 12
  * Descriptive analysis
  * Cross table baseline vs week 12; McNemar Bowker (0) = None
    1. = Trace
    2. = Mild
    3. = Moderate
    4. = Severe

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinik für Klinische Pharmakologie, Allgemeines Krankenhaus Wien, Vienna, Austria